CLINICAL TRIAL: NCT00973466
Title: Prevalence of Asymptomatic and Symptomatic Infection of N. Gonorrheae and C. Trachomatis and Seroprevalence of HSV Typ 2 and Sexual Health Seeking Behaviour in People With HIV Infection in Bern
Brief Title: Prevalence of Sexually Transmitted Infections (STIs) in HIV-infected Patients
Acronym: CTNG
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Pfizer (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Hansjakob Furrer, Leitender Arzt, University Hospital Inselspital, Berne
Other Study IDs: KEK26/09
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: HIV Infections; Neisseria Gonorrhoeae; Chlamydia Trachomatis; Herpes Simplex
Keywords: HIV-infection; Neisseria gonorrhea; Chlamydia trachomatis; Herpes simplex virus; prevalence
MeSH Terms: conditions — HIV Infections; Herpes Simplex; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-infection: All HIV-infected patients attending the Clinic for Infectious Diseases at Berne university hospital, having been sexually active during the past 12 months and having given written informed consent

SUMMARY:
There has been an increase in incidence in sexually transmitted infections in HIV infected patients in the last years. In this study the investigators will prospectively evaluate the prevalence of symptomatic and asymptomatic infections with N. gonorrhea and Ch. trachomatis as well as the seroprevalence of Herpes simplex Type 2 infection in HIV-infected patients attending the clinic for infectious diseases at the Berne University Hospital. In addition, participants will be asked to fill out a questionnaire on sexual behaviour and sexual health.

Study hypothesis: STI prevalence is high in certain risk-groups to justify screening in regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection
* Attending the Clinic for Infectious Diseases from May 09 to November 09
* Sexually active during the last 12 months
* Written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive HIV-infected patients attending the Clinic for Infectious Diseases at Bern University Hospital will be asked to participate in the study if they were sexually active during the last 12 months
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of infection with C.trachomatis, N. gonorrhea and Seroprevalence of HSV 2 infection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hansjakob Furrer, MD, Principal Investigator — University Hospital Berne
Locations (1):
- Clinic for Infectious Diseases, Berne University Hospital, Bern, Switzerland